CLINICAL TRIAL: NCT02965287
Title: Blind Validation of a Metabolomics Based Test for the Non-invasive Screening of Fetal Malformations
Brief Title: Validation of a Test for Fetal Malformations
Status: Completed | Type: Observational
Sponsor: Theoreo Srl (Industry)
Collaborators: Auckland UniServices Ltd. (Industry); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MV-01
Record Dates: First submitted 2016-11-14; First posted 2016-11-16 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2017-10

CONDITIONS: Fetal Anomaly
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 19-21 weeks' gestation: The test validation will be performed on the 1943 serum samples of pregnant women at 19-21 weeks' gestation recruited in New Zealand for the SCOPE Study.
  All the samples will be analyzed to extract and purify the whole metabolome. Metabolites will be characterized through mass spectrometric techniques. These data will be interpreted by means of a bioinformatic algorithm specifically designed for this purpose.
  Interventions: Other: Serum metabolomics profiling
- 14-16 weeks' gestation: Five hundred subjects at 14-16 weeks gestation were randomly selected from the whole cohort of patients. The serum samples collected at 14-16 weeks gestation will be used to test the diagnostic performance at this earlier gestational phase.
  Interventions: Other: Serum metabolomics profiling

INTERVENTIONS:
Other: Serum metabolomics profiling — The serum samples will be used to get a metabolomic profile

SUMMARY:
The investigators have developed a diagnostic test for the evaluation of the presence of fetal malformations through metabolomic analysis of maternal peripheral blood serum by chromatographic techniques and mass spectrometry, and subsequent mathematical modeling analysis of the data by means of multivariate mathematical models specifically developed for this purpose. The study aims at determining the performance parameters (specificity, sensibility, positive predictive value (PPN), negative predictive value (NPV), etc.) of the test and its applicability. To do this, the investigators will use the serum samples of the patients enrolled in New Zealand in the SCOPE Study (www.scopestudy.net), an international study conducted between years 2004-2008.

DETAILED DESCRIPTION:
The test has been developed in a case-control study. In this clinical trial the investigators will test it in a large cohort that is likely to resemble a real population. The purpose of validation is to see if the test is able to recognize the few malformed fetuses in the entire population and especially its specificity in real conditions. In addition, the investigators will check whether particular maternal conditions (such as preeclampsia, gestational diabetes, etc.) or fetal conditions (Small for gestational age, Large for gestational age, etc.) affect the test results.

ELIGIBILITY:
Inclusion criteria were the ones designed by SCOPE Study:

- Nulliparous women, with a singleton pregnancy, between 14wks, 0 days and 16wks, 6 days gestation who give informed consent to participate in SCOPE.

Exclusion criteria were the ones designed by SCOPE Study:

* Unsure of last menstrual period (LMP)
* Unwilling to have ultrasound scan at ≤20 weeks
* ≥3 miscarriages
* ≥3 terminations
* Essential hypertension treated pre-pregnancy
* Moderate-severe hypertension at booking ≥160/100 mmHg
* Diabetes
* Renal disease
* Systemic lupus erythematosus
* Anti-phospholipid syndrome
* Sickle cell disease
* HIV positive
* Major uterine anomaly
* Cervical suture
* Knife cone biopsy
* Ruptured membranes now
* Long term steroids
* Treatment low-dose aspirin
* Treatment calcium (>1g/24h)
* Treatment eicosapentanoic acid (fish oil)
* Treatment vitamin C ≥1000 mg & Vit E ≥400 iu
* Treatment heparin/low molecular weight heparin

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population is the ones selected by the SCOPE Study in New Zealand
Sampling Method: Non-Probability Sample
Enrollment: 1943 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic test performance evaluation in dichotomic classification at 19-21 weeks' gestation | 6 months
  Assessment of the sensitivity, likelihood ratios and performances (diagnostic accuracy) in the identification of a malformed fetus through the analysis of a serum sample from a mother at 19-21 weeks' gestation
Diagnostic test performance evaluation in the individuation of the exact diagnosis of fetal malformation at 19-21 weeks' gestation | 6 months
  Assessment of the sensitivity, likelihood ratios and performances (diagnostic accuracy) in the identification of the type of malformation through the analysis of a serum sample from a mother at 19-21 weeks' gestation

SECONDARY OUTCOMES:
Diagnostic test performance evaluation in dichotomic classification at 14-16 weeks gestation | 6 months
  Assessment of the sensitivity, likelihood ratios and performances (diagnostic accuracy) in the identification of a malformed fetus through the analysis of a serum sample from a mother at 19-21 weeks' gestation
Diagnostic test performance evaluation in the individuation of the exact diagnosis of fetal malformation at 14-16 weeks gestation | 6 months
  Assessment of the sensitivity, likelihood ratios and performances (diagnostic accuracy) in the identification of the type of malformation through the analysis of a serum sample from a mother at 14-16 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Jacopo Troisi, Dr., Principal Investigator — CEO
Locations (1):
- Theoreo srl, Montecorvino Pugliano, Salerno, Italy

IPD SHARING:
Plan to Share IPD: Yes
Test validation of the screening technique will be conducted blinded. The investigators will have access only to the serum samples identified by their unique ID. At the end of the analytical phase, the database containing results will be locked. The database will be transferred to an independent investigator (Prof. Alessio Fasano at Mass General Hospital for Children, Boston, USA) for data analysis. At the same time, information related to pregnancy outcomes (in terms of presence or absence of fetal anomaly) will be transferred from the University of Auckland to the Mass General Hospital for Children, which will provide the blind break and will procced to the estimation of the test performance.

REFERENCES:
- [Background] McCowan LM, Thompson JM, Taylor RS, North RA, Poston L, Baker PN, Myers J, Roberts CT, Dekker GA, Simpson NA, Walker JJ, Kenny LC; SCOPE Consortium. Clinical prediction in early pregnancy of infants small for gestational age by customised birthweight centiles: findings from a healthy nulliparous cohort. PLoS One. 2013 Aug 5;8(8):e70917. doi: 10.1371/journal.pone.0070917. Print 2013. PMID 23940665